CLINICAL TRIAL: NCT01853254
Title: An Open-label, Multicenter Protocol Providing Pegylated Interferon Alfa-2a (Pegasys®) as Monotherapy or in Combination With Ribavirin (Copegus®) for Patients With Chronic Hepatitis C Who Have Participated in Previous Roche or Roche Partner Protocols
Brief Title: A Study of Pegasys (Peginterferon Alfa-2a) Administered Alone or in Combination With Copegus (Ribavirin) in Patients With Chronic Hepatitis C Who Have Participated in Previous Pegasys Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV17590
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- Peginterferon alfa-2a monotherapy or combined with ribavirin (Experimental): The treating investigator decided the most appropriate treatment. It was recommended that participants receive combination therapy.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Both combination and monotherapy for both genotype 2/3 and genotype non-2/3: 180 μg subcutaneously once weekly.
  Other Names: Pegasys
Drug: Ribavirin — For genotype 2/3, 800 mg orally daily, in 2 split doses for 24 weeks. For genotype non-2/3, 1000 mg orally daily for participants weighing < 75 kg or 1200 mg orally daily for participants weighing ≥ 75 kg, in 2 split doses, for 48 weeks.
  Other Names: Copegus

SUMMARY:
This open-label, non-randomized, single arm study will provide treatment or re-treatment with Pegasys (peginterferon alfa-2a) as monotherapy or in combination with Copegus (ribavirin) to patients with chronic hepatitis C infection. Patients who have received prior Pegasys monotherapy or combination therapy or who were considered eligible for treatment with Pegasys in previous donor protocols will be eligible to participate in this study. Treatment will be on investigator's decision according to the approved label for up to 48 weeks, with a 24-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Chronic hepatitis C.
* Compensated liver disease (Child-Pugh Class A).
* Previous participation in a donor protocol in which treatment or re-treatment with Pegasys alone or in combination with Copegus was recommended or deemed appropriate after study completion.
* Have completed safety and efficacy assessments as defined in the donor protocol without violation or any major deviation.
* Have not received any other anti-hepatitis C virus treatment after the completion of the donor protocol.
* For females of childbearing potential, a negative pregnancy test within 24 hours prior to first dose of study drug.
* Fertile patients (male and female) must use 2 reliable forms of contraception (combined) for the duration of the study (treatment and follow-up) in accordance with the locally approved label for Copegus.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Male partners of women who are pregnant.
* Patients with hemoglobinopathies.
* Hepatic decompensation (Child-Pugh Class B or C) before or during treatment.
* Non-responder patients (defined as patients previously treated with Pegasys and Copegus combination therapy at standard doses for at least 12 weeks who did not achieve at least a 2-log drop from their baseline viral load).
* Liver disease other than chronic hepatitis C, including hepatic carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2003-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (60):
- United States (44):
  - Birmingham, Alabama
  - La Jolla, California
  - Long Beach, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Framingham, Massachusetts
  - Worcester, Massachusetts
  - Plymouth, Minnesota
  - Newark, New Jersey
  - Vineland, New Jersey
  - Binghamton, New York
  - Manhasset, New York
  - New York, New York
  - Poughkeepsie, New York
  - Durham, North Carolina
  - Statesville, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Tacoma, Washington
- Australia (2):
  - Adelaide
  - Herston
- Brazil (3):
  - Ribeirão Preto
  - Salvador
  - São Paulo
- Vandœuvre-lès-Nancy, France
- Thessaloniki, Greece
- Italy (2):
  - Bergamo
  - Napoli
- Warsaw, Poland
- Puerto Rico (3):
  - Ponce
  - San Juan
  - Santurce
- Barcelona, Spain
- Taoyuan District, Taiwan
- Plymouth, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin
Started | 272
Completed | 168
Not Completed | 104
Not completed — Abnormal Laboratory Test | 1
Not completed — Adverse Event/Intercurrent Illness | 3
Not completed — Death | 1
Not completed — Failure to Return | 43
Not completed — Insufficient Therapeutic Response | 22
Not completed — Refusal of Treatment | 1
Not completed — Other Protocol Violation | 1
Not completed — Withdrawal of Consent | 16
Not completed — Administrative/Other | 16

BASELINE CHARACTERISTICS:
Arm/Group | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin
Number analyzed (Participants) | 272
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 182
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 24
  Caucasian | 189
  Oriental | 6
  Other | 53
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 172.4 (10.22)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 85.72 (19.803)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event
Time Frame: From Baseline to the end of the study (up to 72 weeks)
Population: All participants analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin
Number analyzed (Participants) | 272
Percentage of participants | 38.2

ADVERSE EVENTS:
Description: All participants analysis set.
Arm/Group | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin
Serious Adverse Events (participants affected / at risk) | 17/272
Other Adverse Events (participants affected / at risk) | 39/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin (N=272)
Anemia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Amaurosis fugax (Eye disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Cryptosporidiosis infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Antibiotic resistant Staphylococcus test positive (Investigations) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a Monotherapy or Combined With Ribavirin (N=272)
Anaemia (Blood and lymphatic system disorders) | 21
Neutropenia (Blood and lymphatic system disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.